CLINICAL TRIAL: NCT00155233
Title: Interaction Between Nalbuphine and Morphine in Postoperative PCA for Gynecologic Patients
Brief Title: Interaction Between Nalbuphine and Morphine in PCA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 931002
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2005-11-23 (Estimated); Status verified 2005-06

CONDITIONS: Postoperative Pain
Keywords: analgeisa; postoperatve; side effects
MeSH Terms: conditions — Pain, Postoperative | interventions — Nalbuphine; Morphine

INTERVENTIONS:
Drug: Nalbuphine and morphine

SUMMARY:
1. Nalbuphine is opioid mu receptor antagonist and kappa receptor agonist
2. This study was designed to investigate the interaction between nalbuphine and morphine

DETAILED DESCRIPTION:
1. Nalbuphine is opioid mu receptor antagonist and kappa receptor agonist
2. This study was designed to investigate the interaction between nalbuphine and morphine
3. The analgesic effect and opioid-related side effects will be investigated

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 y/o
2. Female patients of ASA physical status I to III
3. Scheduled for elective abdominal hysterectomy, myomectomy, or excision of ovarian tumor

Exclusion Criteria:

1. Patients with a definite diagnosis of chronic pain syndrome, psychiatric disorders, or drug abuse (include opioids, NSAIDs, sedatives, antidepressants)
2. Intraoperative fentanyl use > 3 μg/kg
3. Patients with definite diagnosis of esophageal reflux syndrome
4. Use of sedatives, antiemetics, or antipruritics within 24 hours before operation
5. Surgery > 4 hours or laparoscopy surgery

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2005-01

PRIMARY OUTCOMES:
analgesic effect

SECONDARY OUTCOMES:
incidence of opioid-related side effects

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Zen Sun, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan